CLINICAL TRIAL: NCT01309984
Title: An Open-label, Single Initial-dose, Multi-center Study to Assess the Transfer of Fospropofol and Its Active Metabolite, Propofol, to Breast Milk Following Administration of LUSEDRA to Lactating Women Undergoing a Needed Procedure
Brief Title: A Study to Assess the Transfer of Fospropofol and Its Active Metabolite, Propofol, to Breast Milk Following Administration of LUSEDRA to Lactating Women Undergoing a Needed Procedure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2083-A001-405
Record Dates: First submitted 2011-03-02; First posted 2011-03-07 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Lactating Women
Keywords: Monitored anesthesia care
MeSH Terms: interventions — fospropofol; Propofol

ARMS (2):
- arm 1 (Active Comparator)
  Interventions: Drug: Lusedra
- arm 2 (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Lusedra — Pretreatment Phase - approximately 3 hours (Baseline) • Treatment Phase - approximately 8 days (includes Treatment, Discharge [up to 24 hours], and Follow-up Telephone Call on Day 8 post-dose after Discharge)
  Arms: arm 1
Drug: Propofol — Pretreatment Phase - approximately 3 hours (Baseline) • Treatment Phase - approximately 8 days (includes Treatment, Discharge [up to 24 hours], and Follow-up Telephone Call on Day 8 post-dose after Discharge)
  Arms: arm 2

SUMMARY:
The purpose of this study is to assess the transfer of fospropofol and its active metabolite, propofol, to breast milk following administration of LUSEDRA® to lactating women undergoing a needed procedure.

DETAILED DESCRIPTION:
E2083, or LUSEDRA® (fospropofol disodium) Injection, is an intravenous (IV) sedative-hypnotic agent indicated for monitored anesthesia care (MAC) sedation in adult patients undergoing diagnostic or therapeutic procedures.1 It is a water-soluble, phosphono-O-methyl prodrug of propofol. Upon IV injection, the inactive fospropofol undergoes metabolism, most notably by alkaline phosphatase enzymes, to yield the active metabolite (propofol), phosphate, and formaldehyde. Formaldehyde is quickly converted to formate in vivo, and formate is further metabolized by a folate-dependent mechanism.

ELIGIBILITY:
Inclusions:

* Lactating women undergoing a needed procedure expected to last between approximately 10 to 45 minutes
* Subjects should be between 6 weeks and 8 months postpartum
* Lactation must be well-established in subjects
* Subject's infants must be full term and able to bottle-feed
* Infants should be predominantly breast milk fed and should not receive more than one bottle of formula per day

Exclusions:

* Subjects who are pregnant
* Subjects undergoing a breast procedure (eg, biopsy, abscess drainage, etc.)
* Subjects who are not willing to temporarily refrain from nursing their children during the 0-24 hour breast milk collection interval.

(Subjects may resume nursing following this interval).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Total amount (Ae0-24) of propofol transferred to breast milk in 24 hours. | 24 hours
Total amount (Ae0-24) of fospropofol transferred to breast milk in 24 hours | 24 hours
The fraction (%) of the maternal dose transferred to breast milk in 24 hours | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christa Nagy, Study Director — Eisai Inc.
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States